CLINICAL TRIAL: NCT06453135
Title: A Single Center, Open-label, Single-arm Study to Determine the Safety and Efficacy of a Single Dosing Regimen Eculizumab for Prevention of Antibody-Mediated Rejection (AMR) in ABO Blood Group Incompatible Living Donor Kidney Transplantation (ABOi-LDKTx)
Brief Title: Eculizumab for Prevention of Antibody-Mediated Rejection in ABO-Incompatible Living Donor Kidney Transplantation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tao Lin (Other)
Responsible Party: Sponsor-Investigator, Tao Lin, Principal Investigator (PI), West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WestChina-ECU-KT
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Eculizumab; Antibody-mediated rejection
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): A single dose of eculizumab was given on the Day 0 before the transplant surgery.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — On the Day 0, participants received a single dose of eculizumab before the transplant surgery: 900 mg (blood type antibody titer ≥ 1:64 and/or body weight ≥ 60 kg) or 600 mg (blood type antibody titer < 1:64 and body weight < 60 kg). Plasmapheresis was not planned. When participants developed AMR, they may receive additional dose of eculizumab.
  Other Names: Soliris

SUMMARY:
The aim of this study is to determine whether a single dose of eculizumab can effectively prevent antibody-mediated rejection in recipients undergoing living donor kidney transplantation with a different ABO blood group type than their donors

DETAILED DESCRIPTION:
Kidney transplantation is considered the best therapy for patients with end-stage renal disease. ABO-incompatible living donor kidney transplantation (ABOi-LDKTx) is one of the strategies to expand the pool of donors. However, the blood group antibodies in recipients can lead to acute rejection, resulting in transplant failure. Before transplantation, the use of rituximab (RTX) to remove B cells; plasmapheresis to eliminate blood group antibodies can mitigate the occurrence of acute rejection and enhance the success rate of transplantation.

The complement system plays a vital role in antibody-mediated rejection (AMR). Eculizumab can target the C5 protein of the complement system and then block the activation. Therefore, we hypothesize that the pretransplant use of eculizumab may prevent the AMR in ABOi-LDKTx.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years, male or female
2. Suffering from end-stage renal disease and planning for ABO blood group incompatible living donor kidney transplantation
3. Vaccinated against Neisseria meningitides (quadrivalent vaccine), Pneumococcus or H. influenzae at least two weeks prior to using eculizumab
4. Be able to understand the informed consent form and willing to comply with the protocol

Exclusion Criteria:

1. Previous splenectomy
2. Any active bacterial or other infection
3. Known or suspected hereditary complement deficiency
4. Known hypersensitivity to the treatment drug or any of its excipients
5. History of Neisseria meningitidis
6. Any health condition that the investigator believes may interfere with the patient's participation, pose additional risks to the patient, or confound with the patient's assessment (e.g. severe cardiovascular or pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of AMR within 6 months after transplantation | 6 months after kidney transplant surgery

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No